CLINICAL TRIAL: NCT03709953
Title: Efficacy and Safety of Apatinib as Third-line Therapy for Primary Pulmonary Lymphoepithelioid Carcinoma
Acronym: Spark-AL003
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangzhou Institute of Respiratory Disease (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Zhou Chengzhi, Director, Head of pneumology department, Principal Investigator, Clinical Professor, Guangzhou Institute of Respiratory Disease
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Spark-AL003
Record Dates: First submitted 2018-10-11; First posted 2018-10-17 (Actual); Last update posted 2018-10-24 (Actual); Status verified 2018-10

CONDITIONS: Lung Carcinoma
Keywords: apatinib; pulmonary lymphoepithelioid carcinoma
MeSH Terms: conditions — Lung Neoplasms | interventions — apatinib

STUDY DESIGN:
Intervention Model Description: apatinib monotherapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- apatinib (Experimental): apatinib, 500 mg, po, QD; 28 days every cycle
  Interventions: Drug: Apatinib

INTERVENTIONS:
Drug: Apatinib — 500 mg，po，QD； 28 days every cycle
  Other Names: Apatinib mesylate

SUMMARY:
Currently, there is no standard treatment for primary pulmonary lymphoepithelioid carcinoma. Apatinib is a new kind of Vascular endothelial growth factor receptor-2 (VEGFR-2) tyrosine kinase inhibitors (TKIs). A disease-control rate of 75% was found in lung cancer patients in a phase II clinical study. Therefore, researchers hope to explore the efficacy and safety of apatinib in the treatment of primary pulmonary lymphoepithelioid carcinoma.

DETAILED DESCRIPTION:
This study is a prospective, exploratory clinical trial. The purpose of this study was to evaluate the efficacy and safety of apatinib monotherapy in the treatment of primary pulmonary lymphoepithelioid carcinoma.

Thirty-three cases of pulmonary lymphoepithelioid carcinoma were enrolled in this study.

The primary endpoint was median progression-free survival.

ELIGIBILITY:
Inclusion Criteria:

* patients aged from 18 to 75;
* ECOG PS: 0 ~ 2 points;
* lung lymphoepithelioid carcinoma;
* Inoperable stage IV or stage III-B patients who had undergone second-line chemotherapy and had a measurable lesion (according to the RECIST 1.1 standard, the long diameter of the tumor lesion was 10mm in CT scan, the short diameter of the lymph node lesion was 15mm in CT scan, and the lesion was measured without local treatment such as radiotherapy and freezing).
* Life expectancy ≥3 months;
* the main organs are functioning normally:

  1. HB≥80 g/L(no blood transfusion within 14 days); ANC≥1.5×109 /L； PLT≥100×109 /L； WBC≥3×109 /L；
  2. TBIL≤1.5×ULN (upper limit of normal value); ALT and AST ≤2.5×ULN；
  3. creatinine ≤ 1.25 ULN; The clearance rate of creatinine ≥ 60mL/min.
  4. 24-hour urinary protein quantification < 1.0g;
* women of reproductive age (15 to 49 years old) must undergo a urinary pregnancy test within 7 days before starting treatment and the results must be negative. Women are willing to use appropriate methods of contraception;
* Subjects signed the informed consent voluntarily.

Exclusion Criteria:

* Histologically proved to be other types of lung cancer, patients with nasopharyngeal lymphatic epithelial carcinoma with lung metastasis should be excluded.
* Imperfection of upper gastrointestinal physiology, or absorption disorder syndrome, or inability to tolerate oral drugs, or active peptic ulcer;
* Participated in other clinical trials within 4 weeks before the start of the study;
* patients with hypertension who cannot control well through single antihypertensive medication (systolic blood pressure > 140mmhg, diastolic blood pressure > 90mmhg), myocardial ischemia or myocardial infarction, arrhythmia (including QT interval > 440 ms) or cardiac insufficiency;
* Allergic to any ingredient in the drug;
* Patients with abnormal coagulation function, receiving thrombolysis or anticoagulation therapy, bleeding tendency or have clear gastrointestinal bleeding concerns;
* Hyperactive/venous thrombosis events, such as cerebrovascular accident (including transient ischemic attack), deep venous thrombosis and pulmonary embolism occurred in 6 months before the start of the study;
* Wound or fracture has not been healed for a long time;
* urinary protein was greater than ++ and 24-hour urinary protein quantification >1.0 g.
* Severe or uncontrolled infections;
* Substance abuse or mental disorder;
* Objective evidence of a history of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radioactive pneumonia, drug-related pneumonia, and severe impairment of pulmonary function;
* Immunodeficiency, including being HIV-positive, or having other acquired, congenital immunodeficiency diseases, or having a history of organ transplantation;
* Other malignant tumors within 5 years, except cured basal cell carcinoma of the skin and orthotopic carcinoma of the cervix;
* Who have received VEGFR inhibitors, such as sorafenib and sunitinib, etc.;
* pregnant or lactating women;
* the researchers considered it unsuitable for inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2018-10-19 (Actual); Primary Completion 2021-03-31 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
PFS | 24 months
  Median progression-free survival

SECONDARY OUTCOMES:
OS | 24 months
  Median overall survival
ORR | 24 months
  Objective Response Rate
DCR | 24 months
  Disease control rate

OTHER OUTCOMES:
KPS | 24 months
  Karnofsky Performance Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Zhou Chengzhi, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
Update after discussion

REFERENCES:
- [Background] Begin LR, Eskandari J, Joncas J, Panasci L. Epstein-Barr virus related lymphoepithelioma-like carcinoma of lung. J Surg Oncol. 1987 Dec;36(4):280-3. doi: 10.1002/jso.2930360413. PMID 2826922
- [Background] Ngan RK, Yip TT, Cheng WW, Chan JK, Cho WC, Ma VW, Wan KK, Au JS, Law CK. Clinical role of circulating Epstein-Barr virus DNA as a tumor marker in lymphoepithelioma-like carcinoma of the lung. Ann N Y Acad Sci. 2004 Jun;1022:263-70. doi: 10.1196/annals.1318.041. PMID 15251971
- [Background] Lin L, Lin T, Zeng B. Primary lymphoepithelioma-like carcinoma of the lung: An unusual cancer and clinical outcomes of 14 patients. Oncol Lett. 2017 Sep;14(3):3110-3116. doi: 10.3892/ol.2017.6510. Epub 2017 Jun 30. PMID 28928848
- [Background] Kim C, Rajan A, DeBrito PA, Giaccone G. Metastatic lymphoepithelioma-like carcinoma of the lung treated with nivolumab: a case report and focused review of literature. Transl Lung Cancer Res. 2016 Dec;5(6):720-726. doi: 10.21037/tlcr.2016.11.06. PMID 28149767
- [Background] Khokhar N, Nasir H, Amir M, Hassan S, Khan K, Ahmed M. Lymphoepithelioma-Like Carcinoma of the Esophagus: A Rare Tumor. J Coll Physicians Surg Pak. 2017 Sep;27(9):S114-S116. PMID 28969745
- [Background] Lin CY, Chen YJ, Hsieh MH, Wang CW, Fang YF. Advanced primary pulmonary lymphoepithelioma-like carcinoma: clinical manifestations, treatment, and outcome. J Thorac Dis. 2017 Jan;9(1):123-128. doi: 10.21037/jtd.2017.01.25. PMID 28203414
- [Background] Ooi GC, Ho JC, Khong PL, Wong MP, Lam WK, Tsang KW. Computed tomography characteristics of advanced primary pulmonary lymphoepithelioma-like carcinoma. Eur Radiol. 2003 Mar;13(3):522-6. doi: 10.1007/s00330-002-1535-7. Epub 2002 Jul 16. PMID 12594554
- [Background] Mo Y, Shen J, Zhang Y, Zheng L, Gao F, Liu L, Xie C. Primary lymphoepithelioma-like carcinoma of the lung: distinct computed tomography features and associated clinical outcomes. J Thorac Imaging. 2014 Jul;29(4):246-51. doi: 10.1097/RTI.0000000000000070. PMID 24463405
- [Background] Ma H, Wu Y, Lin Y, Cai Q, Ma G, Liang Y. Computed tomography characteristics of primary pulmonary lymphoepithelioma-like carcinoma in 41 patients. Eur J Radiol. 2013 Aug;82(8):1343-6. doi: 10.1016/j.ejrad.2013.02.006. Epub 2013 Mar 5. PMID 23465736
- [Background] Tian S, Quan H, Xie C, Guo H, Lu F, Xu Y, Li J, Lou L. YN968D1 is a novel and selective inhibitor of vascular endothelial growth factor receptor-2 tyrosine kinase with potent activity in vitro and in vivo. Cancer Sci. 2011 Jul;102(7):1374-80. doi: 10.1111/j.1349-7006.2011.01939.x. Epub 2011 May 9. PMID 21443688
- [Background] Jeong JH, Nguyen HK, Lee JE, Suh W. Therapeutic effect of apatinib-loaded nanoparticles on diabetes-induced retinal vascular leakage. Int J Nanomedicine. 2016 Jul 7;11:3101-9. doi: 10.2147/IJN.S108452. eCollection 2016. PMID 27462154
- [Background] Mi YJ, Liang YJ, Huang HB, Zhao HY, Wu CP, Wang F, Tao LY, Zhang CZ, Dai CL, Tiwari AK, Ma XX, To KK, Ambudkar SV, Chen ZS, Fu LW. Apatinib (YN968D1) reverses multidrug resistance by inhibiting the efflux function of multiple ATP-binding cassette transporters. Cancer Res. 2010 Oct 15;70(20):7981-91. doi: 10.1158/0008-5472.CAN-10-0111. Epub 2010 Sep 28. PMID 20876799
- [Background] Tong XZ, Wang F, Liang S, Zhang X, He JH, Chen XG, Liang YJ, Mi YJ, To KK, Fu LW. Apatinib (YN968D1) enhances the efficacy of conventional chemotherapeutical drugs in side population cells and ABCB1-overexpressing leukemia cells. Biochem Pharmacol. 2012 Mar 1;83(5):586-97. doi: 10.1016/j.bcp.2011.12.007. Epub 2011 Dec 16. PMID 22212563
- [Background] Song Z, Yu X, Lou G, Shi X, Zhang Y. Salvage treatment with apatinib for advanced non-small-cell lung cancer. Onco Targets Ther. 2017 Mar 23;10:1821-1825. doi: 10.2147/OTT.S113435. eCollection 2017. PMID 28367065